CLINICAL TRIAL: NCT01465997
Title: A Multicenter, Double-blind, Double-dummy, Follow up Study Evaluating the Long-term Safety of Lacosamide in Comparison With Controlled-release Carbamazepine Used as Monotherapy in Subjects With Partial-onset or Generalized Tonic-clonic Seizures ≥16 Years of Age Coming From the SP0993 Study.
Brief Title: Evaluating Long Term Safety of Lacosamide (LCM) to Carbamazepine Controlled-release (CBZ-CR); Initial Monotherapy in Epilepsy Subjects 16 Years and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB BIOSCIENCES GmbH (Industry)
Collaborators: Eden Sarl (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SP0994; 2010-021238-74 (EudraCT Number)
Expanded Access: NCT03559673 (No longer available)
Record Dates: First submitted 2011-11-02; First posted 2011-11-07 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2017-09

CONDITIONS: Epilepsy; Monotherapy
Keywords: Lacosamide
MeSH Terms: conditions — Epilepsy | interventions — Lacosamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lacosamide (Experimental): 50 and 100 mg tablets of Lacosamide given as 100 mg/day, 200 mg/day, 300 mg/day, 400 mg/day, 500 mg/day or 600 mg/day throughout the Treatment Period (Maximum 3.5 Years)
  Interventions: Drug: Lacosamide
- Carbamazepine-Controlled Release (CBZ-CR) (Active Comparator): 200 mg tablets of Carbamazepine-CR given as 200 mg/day, 400 mg/day, 600 mg/day, 800 mg/day, 1000 mg/day or 1200 mg/day throughout the Treatment Period (Maximum of 3.5 Years)
  Interventions: Drug: Carbamazepine-Controlled Release (CBZ-CR)

INTERVENTIONS:
Drug: Lacosamide — 50 and 100 mg tablets of Lacosamide given as 100 mg/day, 200 mg/day, 300 mg/day, 400 mg/day, 500 mg/day or 600 mg/day throughout the Treatment Period (Maximum 3.5 Years)
  Other Names: VIMPAT film-coated tablets
  Arms: Lacosamide
Drug: Carbamazepine-Controlled Release (CBZ-CR) — 200 mg tablets of Carbamazepine-CR given as 200 mg/day, 400 mg/day, 600 mg/day, 800 mg/day, 1000 mg/day or 1200 mg/day throughout the Treatment Period (Maximum 3.5 Years)
  Other Names: Tegretol® Retard Tablets 200 mg
  Arms: Carbamazepine-Controlled Release (CBZ-CR)

SUMMARY:
Compare safety of Lacosamide (LCM) to Carbamazepine Controlled-Release (CBZ-CR) as monotherapy in newly or recently newly diagnosed subjects with primary safety variables including spontaneous reports of Adverse Events (AEs), withdrawal of subjects due to AEs, reporting of Serious AEs (SAEs).

ELIGIBILITY:
Inclusion Criteria:

* Subject/legal representative is considered reliable and capable of adhering to the protocol
* Subject has remained seizure free and completed the Maintenance Phase of the SP0993; or subject has experienced 1 or more seizures on the first or second target dose during the SP0993 Maintenance Phase
* Subject is expected to benefit from participation in SP0994 in the opinion of the investigator

Exclusion Criteria:

* Subject is receiving any investigational drugs or using any experimental devices in addition to LCM or CBZ-CR
* Subject experienced a seizure at the third target dose during the Evaluation Phase or Maintenance Phase of the SP0993 study
* Subject is taking benzodiazepines for a non-epilepsy indication
* Subject meets a withdrawal criterion from the previous study SP0993
* Subject is experiencing an ongoing SAE from the previous study SP0993
* Subject has a lifetime history of suicide attempt (including an active attempt, interrupted attempt, or aborted attempt), or has suicidal ideation in the past 6 months as indicated by a positive response (Yes) to either Question 4 or Question 5 of the Columbia Suicide Severity Rating Scale (C-SSRS) at Screening. Or subject has a positive response (Yes) to either Question 4 or Question 5 of the C-SSRS at Screening in the "Since Last Visit" version

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 551 (Actual)
Dates: Start 2012-05; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 877 822 9493 (UCB)
Locations (150):
- United States (9):
  - 786, Alabaster, Alabama
  - 799, Huntsville, Alabama
  - 777, Little Rock, Arkansas
  - 789, Panama City, Florida
  - 776, Port Charlotte, Florida
  - 873, Raleigh, North Carolina
  - 794, Oklahoma City, Oklahoma
  - 881, Mansfield, Texas
  - 790, Madison, Wisconsin
- Australia (7):
  - 104, Chatswood
  - 105, Clayton
  - 106, East Gosford
  - 101, Fitzroy
  - 108, Heidelberg
  - 103, Herston
  - 109, Randwick
- Belgium (4):
  - 127, Bruges
  - 134, Bruges
  - 128, Hasselt
  - 126, Leuven
- Bulgaria (6):
  - 805, Blagoevgrad
  - 807, Panagyurishte
  - 803, Pleven
  - 810, Rousse
  - 811, Sofia
  - 809, Veliko Tarnovo
- Canada (4):
  - 152, Greenfield Park
  - 158, Halifax Nova Scotia
  - 156, Hamilton
  - 153, St. John's
- Czechia (5):
  - 185, Brno
  - 190, Ostrava - Vitkovice
  - 184, Prague
  - 189, Prague
  - 180, Zlín
- Finland (2):
  - 205, Helsinki
  - 207, Kuopio
- 236, Nancy, France
- Germany (9):
  - 263, Altenburg
  - 265, Bad Neustadt an der Saale
  - 257, Berlin
  - 262, Berlin
  - 270, Berlin
  - 260, Göttingen
  - 269, Leipzig
  - 256, Marburg
  - 259, Osnabrück
- Greece (3):
  - 495, Ioannina
  - 490, Thessalonikis
  - 493, Thessalonikis
- Hungary (8):
  - 289, Balassagyarmat
  - 283, Budapest
  - 284, Budapest
  - 286, Debrecen
  - 282, Győr
  - 285, Szeged
  - 290, Szekszárd
  - 291, Szombathely
- Italy (5):
  - 310, Bari
  - 309, Modena
  - 308, Padua
  - 314, Prato
  - 311, Roma
- Japan (10):
  - 831, Asaka-shi
  - 833, Hamamatsu
  - 834, Kagoshima
  - 844, Kamakura-shi
  - 843, Miyazaki
  - 835, Nagoya
  - 837, Okayama
  - 828, Saitama-shi
  - 847, Sapporo
  - 832, Shizuoka
- 751, Riga, Latvia
- Lithuania (3):
  - 727, Alytus
  - 724, Kaunas
  - 728, Vilnius
- 547, San Luis Potosí City, Mexico
- Philippines (3):
  - 673, Manila
  - 672, Pasig
  - 676, Quezon City
- Poland (6):
  - 336, Gdansk
  - 340, Katowice
  - 342, Lublin
  - 341, Poznan
  - 338, Szczecin
  - 343, Warsaw
- Portugal (5):
  - 360, Coimbra
  - 362, Lisbon
  - 365, Lisbon
  - 366, Porto
  - 361, Santa Maria da Feira
- Romania (7):
  - 576, Bucharest
  - 569, Cluj-Napoca
  - 570, Iași
  - 579, Iași
  - 571, Sibiu
  - 577, Sibiu
  - 572, Târgu Mureş
- Russia (11):
  - 387, Kazan'
  - 389, Kazan'
  - 396, Kirov
  - 394, Moscow
  - 401, Moscow
  - 390, Nizhny Novgorod
  - 392, Novosibirsk
  - 397, Saint Petersburg
  - 400, Saint Petersburg
  - 386, Smolensk
  - 399, Yaroslavl
- Slovakia (7):
  - 594, Dolný Kubín
  - 598, Dubnica nad Váhom
  - 596, Hlohovec
  - 600, Krompachy
  - 595, Levoča
  - 599, Tornaľa
  - 601, Žilina
- South Korea (8):
  - 525, Busan
  - 521, Daegu
  - 518, Daejeon
  - 517, Seoul
  - 519, Seoul
  - 520, Seoul
  - 523, Seoul
  - 524, Seoul
- Spain (9):
  - 422, Badalona
  - 413, Barcelona
  - 417, Girona
  - 416, Madrid
  - 425, Madrid
  - 419, San Cristóbal de La Laguna
  - 418, San Sebastián
  - 414, Santiago de Compostela
  - 424, Seville
- Sweden (3):
  - 440, Gothenburg
  - 442, Linköping
  - 438, Stockholm
- Switzerland (3):
  - 651, Aarau
  - 654, Biel
  - 653, Lugano
- Thailand (3):
  - 699, Bangkok
  - 702, Bangkok
  - 698, Khon Kaen
- Ukraine (5):
  - 622, Chernihiv
  - 626, Kharkiv
  - 621, Luhansk
  - 625, Odesa
  - 632, Simferopol
- United Kingdom (2):
  - 472, Glasgow
  - 471, Stoke-on-Trent

REFERENCES:
- [Derived] Ben-Menachem E, Dominguez J, Szasz J, Beller C, Howerton C, Jensen L, McClung C, Roebling R, Steiniger-Brach B. Long-term safety and tolerability of lacosamide monotherapy in patients with epilepsy: Results from a multicenter, open-label trial. Epilepsia Open. 2021 Sep;6(3):618-623. doi: 10.1002/epi4.12522. Epub 2021 Aug 2. PMID 34265173
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment started in May 2012 and concluded in January 2017 - 551 patients. Due to the political and civil unrest in Luhansk PAREXEL was not able to conduct further site visits to one site in Ukraine and to collect further data for 2 subjects,they were excluded from SP0994, leaving 549 patients in the Enrolled Set out of 551 initially enrolled.
Pre-assignment Details: A total of 549 subjects gave informed consent in SP0994 and were included in the Enrolled Set, 548 subjects received at least 1 dose of study medication and were included in the Safety Set (SS).
  Participant Flow refers to the Safety Population including all enrolled subjects who received at least 1 dose of study medication in the current study.
Groups:
- Lacosamide: 50 and 100 mg tablets of Lacosamide given as 200 mg/day, 300 mg/day, 400 mg/day, 500 mg/day or 600 mg/day throughout the Treatment Period (Maximum 3.5 Years). CBZ-CR placebo capsules were administered to maintain the blinding.
- Carbamazepine-Controlled Release (CBZ-CR): 200 mg tablets of Carbamazepine-CR given as 400 mg/day, 600 mg/day, 800 mg/day, 1000 mg/day or 1200 mg/day throughout the Treatment Period (Maximum of 3.5 Years). Lacosamide placebo capsules were administered to maintain the blinding.
Period: Overall Study
Arm/Group | Lacosamide | Carbamazepine-Controlled Release (CBZ-CR)
Started | 279 | 269
Completed | 211 | 180
Not Completed | 68 | 89
Not completed — Adverse Event | 12 | 22
Not completed — Lack of Efficacy | 13 | 1
Not completed — Protocol Violation | 1 | 4
Not completed — Lost to Follow-up | 6 | 9
Not completed — Withdrawal by Subject | 32 | 35
Not completed — investigator's decision | 1 | 1
Not completed — Death | 0 | 1
Not completed — sponsor's decision | 1 | 1
Not completed — subject withdrew consent | 1 | 0
Not completed — local lab unblinded site | 1 | 0
Not completed — withdrew before follow-up | 0 | 13
Not completed — decision by site staff | 0 | 1
Not completed — subject left participation SP0993 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis group for Baseline Characteristics is the Safety Set (SS). The SS consists of all subjects in the Enrolled Set who have received at least 1 dose of study medication.
Arm/Group | Lacosamide | Carbamazepine-Controlled Release (CBZ-CR) | Total Title
Number analyzed (Participants) | 279 | 269 | 548
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 8 | 16
  Between 18 and 65 years | 230 | 225 | 455
  >=65 years | 41 | 36 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (17.2) | 42.7 (16.7) | 42.9 (17.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 125 | 250
  Male | 154 | 144 | 298

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With at Least One Treatment-emergent Adverse Event (AE) During the Treatment Phase (Maximum of 3.5 Years)
Description: Treatment-emergent AEs were defined as those events which started on or after the date of first dose of SP0994 study medication, or events in which severity worsened on or after the date of first dose of SP0994 study medication. AEs which occurred within 30 days after last dose of study medication were considered treatment emergent.
Time Frame: Up to 3.5 Years (Duration of the Treatment Phase)
Measure: Count of Participants; unit: Participants
Groups:
- Lacosamide (SS): 50 and 100 mg tablets of Lacosamide given as 200 mg/day, 300 mg/day, 400 mg/day, 500 mg/day or 600 mg/day throughout the Treatment Period (Maximum 3.5 Years). CBZ-CR placebo capsules were administered to maintain the blinding.
- Carbamazepine-Controlled Release (CBZ-CR) (SS): 200 mg tablets of Carbamazepine-CR given as 400 mg/day, 600 mg/day, 800 mg/day, 1000 mg/day or 1200 mg/day throughout the Treatment Period (Maximum of 3.5 Years). Lacosamide placebo capsules were administered to maintain the blinding.
Arm/Group | Lacosamide (SS) | Carbamazepine-Controlled Release (CBZ-CR) (SS)
Number analyzed (Participants) | 279 | 269
Participants | 181 | 182

2. Primary Outcome: Number of Subjects Who Withdrew From the Study Due to a Treatment-emergent Adverse Event (AE) During the Treatment Phase (Maximum 3.5 Years)
Description: as for outcome 1
Time Frame: Up to 3.5 Years (Duration of the Treatment Phase)
Measure: Count of Participants; unit: Participants
Arm/Group | Lacosamide | Carbamazepine-Controlled Release (CBZ-CR)
Number analyzed (Participants) | 279 | 269
Participants | 12 | 21

3. Primary Outcome: Number of Subjects With at Least One Treatment-emergent Serious Adverse Event (SAE) During the Treatment Phase (Maximum of 3.5 Years)
Description: A Serious Adverse Event is any untoward medical occurrence that at any dose results in death, is life threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity is a congenital anomaly/birth defect.
Time Frame: Up to 3.5 Years (Duration of the Treatment Phase)
Measure: Count of Participants; unit: Participants
Arm/Group | Lacosamide | Carbamazepine-Controlled Release (CBZ-CR)
Number analyzed (Participants) | 279 | 269
Participants | 32 | 22

ADVERSE EVENTS:
Time Frame: During the entire study period, up to 5 years
Arm/Group | Lacosamide (SS) | Carbamazepine-Controlled Release (CBZ-CR) (SS)
Serious Adverse Events (participants affected / at risk) | 32/279 | 22/269
Other Adverse Events (participants affected / at risk) | 45/279 | 42/269
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (SS) (N=279) | Carbamazepine-Controlled Release (CBZ-CR) (SS) (N=269)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Vestibular ataxia (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Exophthalmos (Eye disorders) | 0 (0) | 1 (1)
Lumbar hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 3 (4)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
White matter lesion (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Reversible ischaemic neurological deficit (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Pregnancy on contraceptive (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 2 (2)
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Epididymitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (SS) (N=279) | Carbamazepine-Controlled Release (CBZ-CR) (SS) (N=269)
Nasopharyngitis (Infections and infestations) | 20 (40) | 16 (22)
Headache (Nervous system disorders) | 17 (28) | 16 (26)
Dizziness (Nervous system disorders) | 12 (13) | 17 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days